CLINICAL TRIAL: NCT00096122
Title: PHASE I-II STUDY OF IDARUBICIN, CYTARABINE AND R115777 (TIPIFARNIB, ZARNESTRA; 702818; IND 58359), A FARNESYLTRANSFERASE INHIBITOR, IN PATIENTS WITH HIGH-RISK MYELODYSPLASTIC SYNDROMES AND ACUTE MYELOID LEUKEMIAS
Brief Title: Idarubicin, Cytarabine, and Tipifarnib in Treating Patients With Newly Diagnosed Myelodysplastic Syndromes or Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02862; 2003-0563; 6625; N01CM62202 (NIH)
Record Dates: First submitted 2004-11-09; First posted 2004-11-09 (Estimated); Results first posted 2011-07-15 (Estimated); Last update posted 2014-05-26 (Estimated); Status verified 2013-06

CONDITIONS: Adult Acute Basophilic Leukemia; Adult Acute Eosinophilic Leukemia; Adult Acute Megakaryoblastic Leukemia (M7); Adult Acute Minimally Differentiated Myeloid Leukemia (M0); Adult Acute Monoblastic Leukemia (M5a); Adult Acute Monocytic Leukemia (M5b); Adult Acute Myeloblastic Leukemia With Maturation (M2); Adult Acute Myeloblastic Leukemia Without Maturation (M1); Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Acute Myelomonocytic Leukemia (M4); Adult Erythroleukemia (M6a); Adult Pure Erythroid Leukemia (M6b); Childhood Myelodysplastic Syndromes; Chronic Myelomonocytic Leukemia; de Novo Myelodysplastic Syndromes; Refractory Anemia With Excess Blasts; Refractory Anemia With Excess Blasts in Transformation; Secondary Acute Myeloid Leukemia; Secondary Myelodysplastic Syndromes; Untreated Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Basophilic, Acute; Leukemia, Eosinophilic, Acute; Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myeloid, Acute; Congenital Abnormalities; Leukemia, Myelomonocytic, Acute; Leukemia, Erythroblastic, Acute; Leukemia, Myelomonocytic, Chronic; Anemia, Refractory, with Excess of Blasts | interventions — Cytarabine; Idarubicin; tipifarnib

ARMS (1):
- Arm I (Experimental): See Detailed Description
  Interventions: Drug: cytarabine; Drug: idarubicin; Drug: tipifarnib

INTERVENTIONS:
Drug: cytarabine — Given IV
  Other Names: ARA-C; arabinofuranosylcytosine; arabinosylcytosine; Cytosar-U; cytosine arabinoside
Drug: idarubicin — Given IV
  Other Names: 4-demethoxydaunorubicin; 4-DMDR; DMDR; IDA
Drug: tipifarnib — Given orally
  Other Names: R115777; Zarnestra

SUMMARY:
This phase I/II trial is studying the side effects and best dose of tipifarnib when given with idarubicin and cytarabine and to see how well it works in treating patients with newly diagnosed myelodysplastic syndromes or acute myeloid leukemia. Drugs used in chemotherapy, such as idarubicin and cytarabine, work in different ways to stop cancer cells from dividing so they stop growing or die. Tipifarnib (Zarnestra) may stop the growth of cancer cells by blocking the enzymes necessary for their growth. Giving idarubicin and cytarabine with tipifarnib may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the tolerability of the combination of R115777 (Zarnestra™) and Idarubicin plus cytarabine by defining the DLT and MTD. (Phase I) II. To determine the efficacy of the combination of Idarubicin, cytarabine and ZARNESTRA in patients with high-risk MDS and AML. (Phase II)

OUTLINE: This is a dose-escalation study of tipifarnib. Patients are stratified according to age (< 50 versus ≥ 50) and, in patients ≥ 50 years of age, cytogenetics (diploid versus unfavorable).

INDUCTION THERAPY:

PHASE I: Patients receive cytarabine IV continuously on days 1-3 (or 1-4), idarubicin intravenous (IV) over 1 hour on days 1-3, and oral tipifarnib twice daily on days 1-21. Treatment repeats every 21 days for up to 2 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 6 patients receive escalating doses of tipifarnib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.

PHASE II: Patients receive cytarabine, idarubicin, and tipifarnib as in phase I at the MTD.

Patients in both phases who respond to induction therapy proceed to consolidation maintenance therapy.

CONSOLIDATION MAINTENANCE THERAPY: Patients receive consolidation therapy comprising cytarabine IV continuously on days 1-3, idarubicin IV over 1 hour on days 1-2, and tipifarnib twice daily on days 1-14. Treatment repeats every 4-6 weeks for 5 courses in the absence of unacceptable toxicity.

Patients then begin maintenance therapy comprising oral tipifarnib twice daily on day 1-21. Treatment repeats every 4-6 weeks for 6 courses in the absence of unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of 1) AML (WHO classification definition of > 20% blasts), or 2) high risk MDS (defined as the presence of > 10% blasts)
* Patients must be chemo-naïve, i.e. not have received any prior chemotherapy (except hydrea) for AML or MDS; they could have received transfusions, hematopoietic growth factors or vitamins; temporary measures such as pheresis or hydrea (0.5 to 5g daily for up to 3 days) are allowed
* ECOG PS of 0-1 at screening
* Creatinine =< 2 mg/dl
* Total bilirubin =< 2 mg/dL, unless increase is due to hemolysis
* Transaminases (SGPT) =< 2.5 x ULN
* Ability to take oral medication
* Ability to understand and provide signed informed consent

Exclusion Criteria:

* Subjects with APL
* Presence of active systemic infection
* Any coexisting medical condition that in the judgment of the treating physician is likely to interfere with study procedures or results
* Nursing women, women of childbearing potential with positive urine pregnancy test, or women of childbearing potential who are not willing to maintain adequate contraception (such as birth control pills, IUD, diaphragm, abstinence, or condoms by their partner) over the entire course of the study
* Known allergy to imidazole drugs (such as clotrimazole, ketoconazole, miconazole, econazole, fenticonazole, isoconazole, sulconazole, tioconazole, terconazole)

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2004-09; Primary Completion 2006-09 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Cortes, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 9/16/2004 to 9/22/2006. All patients registered at The University of Texas M.D. Anderson Cancer Center.
Pre-assignment Details: One participant enrolled was excluded from the study.
Groups:
- Idarubicin, Cytarabine + Tipifarnib: Cytarabine 1.5 g/m^2 and Idarubicin 12 mg/m^2 intravenous (IV) continuously on days 1-3 (or 1-4), with Oral Tipifarnib 200/300 twice daily on days 1-21, repeats every 21 days.
Period: Overall Study
Arm/Group | Idarubicin, Cytarabine + Tipifarnib
Started | 95
Completed | 95
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Idarubicin, Cytarabine + Tipifarnib
Number analyzed (Participants) | 95
Age, Continuous [Median (Full Range); unit: years] | 50 [17 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53
  Male | 42
Region of Enrollment [Number; unit: participants]
  United States | 95

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Response
Description: Complete Response (CR) is required bone marrow blasts ≤5% and recovery of normal hematopoiesis with an absolute neutrophil count (ANC) of 1*10^9/L or more and platelet count of 100*10^9/L or more; and a complete response without platelets (CRp) is the same criteria as CR but with platelet counts from 20*10^9/L to less than 100*10^9/L.
Time Frame: 21 Day Cycle
Population: Analysis was per protocol.
Measure: Number; unit: Participants
Arm/Group | Idarubicin, Cytarabine + Tipifarnib
Number analyzed (Participants) | 95
Participants
  CR | 61
  CRp | 9

ADVERSE EVENTS:
Time Frame: 5 years 4 months
Arm/Group | Idarubicin, Cytarabine + Tipifarnib
Serious Adverse Events (participants affected / at risk) | 46/95
Other Adverse Events (participants affected / at risk) | 95/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Idarubicin, Cytarabine + Tipifarnib (N=95)
Infection (Infections and infestations) | 12 (14)
Febrile neutropenia (Infections and infestations) | 14 (21)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Hyperbilirubinemia (Hepatobiliary disorders) | 6 (6)
Death (General disorders) | 5 (5)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2)
Enteritis (Gastrointestinal disorders) | 1 (1)
Hemorrhage (Vascular disorders) | 5 (5)
Typhilitis (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Decreased left ventricular ejection fraction (LVEF) (Cardiac disorders) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 2 (2)
Renal Failure (Renal and urinary disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Edema (General disorders) | 1 (1)
Bilateral pleural effusions (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Confusion (Nervous system disorders) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Idarubicin, Cytarabine + Tipifarnib (N=95)
Diarrhea (Gastrointestinal disorders) | 66 (66)
Nausea/Vomiting (Gastrointestinal disorders) | 54 (54)
Rash/Puritis (Skin and subcutaneous tissue disorders) | 51 (51)
Hyperbilirubinemia (Hepatobiliary disorders) | 25 (25)
Mucositis (Gastrointestinal disorders) | 23 (23)
Pain (General disorders) | 27 (27)
Fatigue (General disorders) | 20 (20)
Mood alteration (Nervous system disorders) | 12 (12)
Hypotension (Cardiac disorders) | 12 (12)
Hypokalemia (Metabolism and nutrition disorders) | 12 (12)
Edema (General disorders) | 11 (11)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9 (9)
Constipation (Gastrointestinal disorders) | 11 (11)
Hypoalbuminemia (Metabolism and nutrition disorders) | 10 (10)
Hyperglycemia (Metabolism and nutrition disorders) | 10 (10)
Hypophosphatemia (Metabolism and nutrition disorders) | 8 (8)
Anorexia (Gastrointestinal disorders) | 8 (8)
Elevated creatinine (Renal and urinary disorders) | 7 (7)
Hypocalcemia (Metabolism and nutrition disorders) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less